CLINICAL TRIAL: NCT00318279
Title: Benefits of a Surgical Skills Lab Vascular Anastomosis Simulator: A Randomized Controlled Trial
Brief Title: Evaluation of Surgical Simulator for Practicing a Vascular Anastomosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Dr. M. Quantz, Lawson Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: R-05-826; 11858E
Record Dates: First submitted 2006-04-24; First posted 2006-04-26 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Education, Medical
Keywords: Surgical education; Vascular anastomosis; Simulator; Randomized controlled trial

INTERVENTIONS:
Device: Surgical simulator to practice vascular anastomosis

SUMMARY:
To determine if practicing an aorto-saphenous vein anastomosis on a low-fidelity surgical simulator allows trainees to produce a higher quality anastomosis in a shorter period of time, than a group that only learns by watching a video.

DETAILED DESCRIPTION:
For many years, surgical training has been considered an apprenticeship, where the training experiences of residents, have been in real operative settings on living patients. We propose a study to demonstrate that - a low-fidelity simulation of an aorta-proximal vein graft anastomosis as in heart bypass surgery, using anatomical replicates (a special hydrogel polymer with properties similar to human vascular tissue) - is an effective, low-cost simulator for learning this surgical skill, and will provide the trainee with the ability to perform a better anastomosis in a shorter period of time.

Hypothesis: Practicing an aorto-saphenous vein anastomosis on a low-fidelity surgical simulator will advance the trainees' learning curve. This will allow trainees to produce a higher quality anastomosis in a shorter period of time, than a group that only learns by watching a video and will lead to enhanced patient safety.

ELIGIBILITY:
Inclusion Criteria:

* 1st year surgical resident at The University of Western Ontario
* Anastomosis naive - the subject must not have performed a human vascular anastomosis in the past (it is acceptable if they have observed one being performed in the past)

Exclusion Criteria:

* Completed a human vascular anastomosis as the primary operator/surgeon in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2007-05 (Actual); Study Completion 2007-09

PRIMARY OUTCOMES:
Quality of final vascular anastomosis based on validated scale

SECONDARY OUTCOMES:
Global rating of operative skill based on validated scale (final anastomosis)
Time taken to complete final anastomosis
Time taken to complete initial and final anastomosis (experimental group only)
Anastomotic leakage for final anastomosis
Anastomotic patency for final anastomosis

CONTACTS AND LOCATIONS:
Overall Officials: Mackenzie A Quantz, MD, FRCSC, Principal Investigator — The University of Western Ontario; Pavan K Koka, BSc, MD, Principal Investigator — The University of Western Ontario
Locations (1):
- Kelman Advanced Centre for Learning, The University of Western Ontario, London, Ontario, Canada

REFERENCES:
- [Background] Grober ED, Hamstra SJ, Wanzel KR, Reznick RK, Matsumoto ED, Sidhu RS, Jarvi KA. The educational impact of bench model fidelity on the acquisition of technical skill: the use of clinically relevant outcome measures. Ann Surg. 2004 Aug;240(2):374-81. doi: 10.1097/01.sla.0000133346.07434.30. PMID 15273564
- [Background] Grober ED, Hamstra SJ, Wanzel KR, Reznick RK, Matsumoto ED, Sidhu RS, Jarvi KA. Laboratory based training in urological microsurgery with bench model simulators: a randomized controlled trial evaluating the durability of technical skill. J Urol. 2004 Jul;172(1):378-81. doi: 10.1097/01.ju.0000123824.74075.9c. PMID 15201815
- [Background] Anastakis DJ, Regehr G, Reznick RK, Cusimano M, Murnaghan J, Brown M, Hutchison C. Assessment of technical skills transfer from the bench training model to the human model. Am J Surg. 1999 Feb;177(2):167-70. doi: 10.1016/s0002-9610(98)00327-4. PMID 10204564
- [Background] Hance J, Aggarwal R, Stanbridge R, Blauth C, Munz Y, Darzi A, Pepper J. Objective assessment of technical skills in cardiac surgery. Eur J Cardiothorac Surg. 2005 Jul;28(1):157-62. doi: 10.1016/j.ejcts.2005.03.012. Epub 2005 Apr 9. PMID 15982599
- [Background] Watterson JD, Beiko DT, Kuan JK, Denstedt JD. Randomized prospective blinded study validating acquistion of ureteroscopy skills using computer based virtual reality endourological simulator. J Urol. 2002 Nov;168(5):1928-32. doi: 10.1016/S0022-5347(05)64265-6. PMID 12394678
- [Background] Reznick R, Regehr G, MacRae H, Martin J, McCulloch W. Testing technical skill via an innovative "bench station" examination. Am J Surg. 1997 Mar;173(3):226-30. doi: 10.1016/s0002-9610(97)89597-9. PMID 9124632
- [Background] Youngblood PL, Srivastava S, Curet M, Heinrichs WL, Dev P, Wren SM. Comparison of training on two laparoscopic simulators and assessment of skills transfer to surgical performance. J Am Coll Surg. 2005 Apr;200(4):546-51. doi: 10.1016/j.jamcollsurg.2004.11.011. PMID 15804468
- [Background] Beard JD, Jolly BC, Newble DI, Thomas WE, Donnelly J, Southgate LJ. Assessing the technical skills of surgical trainees. Br J Surg. 2005 Jun;92(6):778-82. doi: 10.1002/bjs.4951. PMID 15810048
- [Background] Clark JA, Volchok JA, Hazey JW, Sadighi PJ, Fanelli RD. Initial experience using an endoscopic simulator to train surgical residents in flexible endoscopy in a community medical center residency program. Curr Surg. 2005 Jan-Feb;62(1):59-63. doi: 10.1016/j.cursur.2004.07.002. PMID 15708148
- [Background] Backstein D, Agnidis Z, Sadhu R, MacRae H. Effectiveness of repeated video feedback in the acquisition of a surgical technical skill. Can J Surg. 2005 Jun;48(3):195-200. PMID 16013622
- [Result] Lachin JM. Introduction to sample size determination and power analysis for clinical trials. Control Clin Trials. 1981 Jun;2(2):93-113. doi: 10.1016/0197-2456(81)90001-5. PMID 7273794